CLINICAL TRIAL: NCT07218913
Title: Phase 1 Trial of Pedmark in Men Receiving Cisplatin for Metastatic Germ Cell Tumor
Brief Title: Testing the Addition of Pedmark to Cisplatin Chemotherapy for Reducing Drug-Induced Ear Damage in Men With Stage II-III Metastatic Testicular Germ Cell Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25407; NCI-2025-07298 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25407 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss; Metastatic Malignant Germ Cell Tumor; Metastatic Malignant Nongerminomatous Germ Cell Tumor; Metastatic Malignant Testicular Non-Seminomatous Germ Cell Tumor; Metastatic Testicular Seminoma; Stage II Testicular Cancer AJCC v8; Stage III Testicular Cancer AJCC v8
MeSH Terms: conditions — Hearing Loss; Seminoma; Testicular Neoplasms | interventions — Hearing; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Magnetic Resonance Spectroscopy; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (SOC cisplatin) (Active Comparator): Patients receive cisplatin IV over 60 minutes on days 1-5 or 2-5 of each SOC cisplatin-based chemotherapy regimen cycle. Cycles repeat every 21 days for 3-4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial.
  Interventions: Procedure: Audiometric Test; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm II (SOC cisplatin, Pedmark) (Experimental): Patients receive cisplatin IV over 60 minutes on days 1-5 or 2-5 of each SOC cisplatin-based chemotherapy regimen cycle. Patients also receive Pedmark IV over 30 minutes, 6 hours after each SOC cisplatin infusion, on days 1-5 or 2-5 of each cycle. Cycles repeat every 21 days for 3-4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial.
  Interventions: Procedure: Audiometric Test; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Sodium Thiosulfate Anhydrous

INTERVENTIONS:
Procedure: Audiometric Test — Ancillary studies
  Other Names: Audiometric Testing; Audiometry; Hearing Test
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Sodium Thiosulfate Anhydrous — Given IV
  Other Names: Disodium Thiosulfate; Sodium Thiosulfate, Anhydrous; Thiosulfuric Acid, Disodium Salt
  Arms: Arm II (SOC cisplatin, Pedmark)

SUMMARY:
This phase I trial evaluates whether adding Pedmark to standard of care cisplatin-based chemotherapy reduces drug-induced ear damage (ototoxicity) in men with stage II-III testicular germ cell tumors that have spread from where they first started (primary site) to other places in the body (metastatic). Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Cisplatin-induced ototoxicity remains a major concern in adult patients with germ cell tumors as nearly four out of five patients develop hearing loss after treatment. Cisplatin is thought to cause ear damage by the production of chemically reactive molecules called reactive oxygen species. These molecules can cause damage when their levels get too high. Pedmark may reduce the negative side effects of cisplatin by neutralizing these reactive molecules. Pedmark has been approved for reducing the risk of cisplatin-induced ototoxicity in pediatric patients and older patients with solid tumors that haven't spread to other parts of the body. Adding Pedmark to cisplatin-based chemotherapy treatment may reduce ototoxicity in adult men with stage I-III testicular metastatic germ cell tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the incidence of clinically meaningful ototoxicity in adults with metastatic germ cell tumor (GCT) receiving sodium thiosulfate anhydrous (Pedmark) plus cisplatin-based chemotherapy compared to those receiving cisplatin-based chemotherapy alone.

SECONDARY OBJECTIVES:

I. Assess the incidence of high-frequency ototoxicity (affecting frequencies within 8000-12,500 Hz) between adults in both arms.

II. Assess the severity and progression of ototoxicity between adults in both arms.

III. Determine the safety and tolerability of Pedmark plus cisplatin-based chemotherapy compared to cisplatin-based chemotherapy alone.

IV. Examine the efficacy of Pedmark plus cisplatin-based chemotherapy compared to cisplatin-based chemotherapy alone.

EXPLORATORY OBJECTIVES:

I. Evaluate the incidence of tinnitus between adults in both arms. II. Disease assessment 6 months post-primary treatment in both arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cisplatin intravenously (IV) over 60 minutes on days 1-5 or 2-5 of each standard of care (SOC) cisplatin-based chemotherapy regimen cycle. Cycles repeat every 21 days for 3-4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the trial.

ARM II: Patients receive cisplatin IV over 60 minutes on days 1-5 or 2-5 of each SOC cisplatin-based chemotherapy regimen cycle. Patients also receive Pedmark IV over 30 minutes, 6 hours after each SOC cisplatin infusion, on days 1-5 or 2-5 of each cycle. Cycles repeat every 21 days for 3-4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the trial.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year and then per SOC for year 2.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Willing and able to sign informed consent form
* Willing and able to participate in baseline and serial audiometry exams
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) of 0 or 1 or Karnofsky score ≥ 70
* Histologically confirmed germ cell tumor (seminoma or non-seminoma)
* Presence of metastatic disease (stage II or III)
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Receiving first or second line cisplatin-based chemotherapy
* Planned cumulative cisplatin dose of ≥ 300mg/m^2 (including previous treatment)
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin ≥ 9g/dL

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 X upper limit of normal (ULN)

  * Patients with known Gilbert disease who have serum bilirubin level < 3 x ULN may be enrolled
* Aspartate aminotransferase (AST) ≤ 3.0 x ULN
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN
* Creatinine clearance of ≥ 60 mL/min per the Cockcroft-Gault formula or serum creatinine ≤ 1.5 x ULN
* * If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN

  * If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* * If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN

  * If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Advise male patients with female partners of reproductive potential to use effective contraception during treatment and for 11 months after the last dose of cisplatin for injection

Exclusion Criteria:

* Any cisplatin-based therapies within 4 weeks prior to initiation of study treatment
* If cisplatin infusion during study is planned to be longer than 6 hours, as Pedmark safety and efficacy has not been established when administered following longer cisplatin infusions
* Chronic steroid use, defined as greater than prednisone 5 mg daily for longer than 21 days (steroids used as antiemetic during treatment is permitted)
* Concurrent use of other ototoxic drugs other than cisplatin (loop diuretics, aminoglycosides, etc)
* Patient must adhere to low sodium diet given other comorbidities
* History of severe hypersensitivity to sodium thiosulfate or any components such as sulfites or thiols
* Known symptomatic brain metastases, leptomeningeal carcinomatosis, or prior cranial irradiation
* Deemed cisplatin ineligible due to poor performance status, cardiac dysfunction, renal insufficiency, or significant peripheral neuropathy
* Greater than or equal to moderate hearing loss (HL) at baseline per World Health Organization (WHO) classification
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Uncontrolled atrial fibrillation or hypertension
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-03-04 (Estimated); Primary Completion 2031-01-22 (Estimated); Study Completion 2031-01-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically meaningful ototoxicity | Up to 6 months post-treatment
  Will compare the proportion of patients who experience clinically meaningful ototoxicity between adults with germ cell tumor (GCT) receiving Pedmark plus cisplatin-based chemotherapy compared to those receiving cisplatin-based chemotherapy alone. Clinically meaningful ototoxicity is defined by a > 20 decibel (dB) threshold shift at a single frequency, a > 10 dB shift at two adjacent frequencies, or a change to "no response" at three consecutive frequencies as long as these frequencies fall between 250-8000 hertz (Hz) which impacts speech understanding. The corresponding 95% confidence interval (CI) will be constructed using the Clopper-Pearson exact method. The proportion of patients who develop clinically meaningful ototoxicity will be compared between arms using a one-sided Fisher's exact test.

SECONDARY OUTCOMES:
Incidence of high-frequency ototoxicity | Up to 6 months post-treatment
  Will compare the proportion of patients who experience high-frequency ototoxicity between adults with GCT receiving Pedmark plus cisplatin-based chemotherapy compared to those receiving cisplatin-based chemotherapy alone. High frequency ototoxicity is defined by a > 20 dB threshold shift at a single frequency, a > 10 dB shift at two adjacent frequencies, or a change to "no response" at three consecutive frequencies as long as these frequencies fall between 8000-12,00 Hz. Will be estimated with 95% CIs by the Clopper-Pearson exact method. The proportion of patients who develop high-frequency ototoxicity will be compared between arms using a one-sided Fisher's exact test.
Degree of ototoxicity | Baseline to 1, 3, and 6 months post-treatment
  Audiometry results between adults with GCT receiving Pedmark plus cisplatin-based chemotherapy will be compared to those receiving cisplatin-based chemotherapy alone. This will be decided by the audiologist per World Health Organization classification. Longitudinal changes in degree of ototoxicity will be summarized descriptively and analyzed using repeated-measures models to compare changes from baseline across time points between treatment arms.
Incidence of adverse events (AEs) | Up to 6 months post-treatment
  Will evaluate the rate of adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 in adults with GCT receiving Pedmark plus cisplatin-based chemotherapy compared to those receiving cisplatin-based chemotherapy alone. The safety evaluation will be based on all patients that received at least one dose of the drug and will include AEs, serious AEs, and changes from baseline in laboratory evaluations, vital signs, and physical examinations. Summaries will be provided overall and by treatment group. The number and percentage of subjects reporting will be summarized overall and by CTCAE grade. All patients will be evaluable for toxicity from the time of their first treatment with cisplatin-based chemotherapy ± Pedmark.
Progression-free survival (PFS) | From start of treatment to time of progressive disease or death, assessed up to 2 years
  Will be assessed per Response Evaluation Criteria in Solid Tumors version 1.1. The difference in PFS between treatment arms will be estimated using the Kaplan-Meier method, with survival curves generated for each group. Statistical comparison of PFS between arms will be conducted using the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chehrazi-Raffle, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States